CLINICAL TRIAL: NCT03597516
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Durability, Safety, and Tolerability of RP-G28 in Patients With Lactose Intolerance
Brief Title: Evaluation of the Efficacy, Durability, Safety, and Tolerability of RP-G28 in Patients With Lactose Intolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ritter Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G28-006
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Lactose Intolerance
Keywords: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — RP-G28

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study conducted in the United States (US). The study is comprised of 4 study periods.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RP-G28 (Experimental): galacto-oligosaccharide, spray-dried powder for reconstitution for oral administration, 7.5 grams 2 times per day
  Interventions: Drug: RP-G28
- Placebos (Placebo Comparator): maltodextrin, powder for reconstitution for oral administration, 7.5 grams 2 times per day
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: RP-G28 — powder for reconstitution for oral administration
  Arms: RP-G28
Drug: Placebos — powder for reconstitution for oral administration
  Arms: Placebos

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study conducted in the United States (US) to assess the efficacy of RP-G28 compared to placebo on symptom reduction related to lactose intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-75 years of age, inclusive, at screening;
* Intolerance to milk and other dairy products;
* Patient agrees to refrain from all other treatments and products used for lactose intolerance, to follow diet modifications required during periods of the study that include abstinence from all dairy in some periods and consuming dairy in other periods;
* Patient meets the defined minimum lactose intolerance symptom composite score; and
* Patient has positive Hydrogen Breath Test (HBT) results for lactase deficiency.

Exclusion Criteria:

* Patient has a disorder associated with abnormal gastrointestinal motility such as gastroparesis (from any cause), amyloidosis, neuromuscular diseases (including Parkinson's disease), collagen vascular diseases, uremia, or malnutrition;
* Patient has undergone bowel preparation for endoscopic or radiologic investigation within 4 weeks of Screening (example, colonoscopy preparation);
* Patient has a history of surgery that alters the normal function of the gastrointestinal tract including, but not limited to: fundoplication, gastrointestinal bypass surgery, bariatric surgery, gastric banding, colostomy, vagotomy, pyloroplasty, colectomy or other surgery for Crohn's disease or ulcerative colitis; and
* Patient has received antibiotic treatment, or had a high colonic enema, colonic irrigation, colonic hydrotherapy, or colonic cleaning within 30 days prior to or during Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the Lactose Intolerance (LI) symptom composite score compared to placebo | Day 61
  Change from baseline of the LI symptom composite score compared to placebo. The LI symptom composite score includes abdominal pain, abdominal bloating, abdominal cramping, and abdominal gas.

SECONDARY OUTCOMES:
Proportion of patients with a meaningful reduction in LI composite score. | Day 61
  Proportion of patients with a meaningful reduction in LI composite score. The LI symptom composite score includes abdominal pain, abdominal bloating, abdominal cramping, and abdominal gas.

CONTACTS AND LOCATIONS:
Overall Officials: Sharron Gargosky, PhD, Study Director — Ritter Pharmceuticals, Inc.
Locations (34):
- United States (34):
  - Research Facility, Birmingham, Alabama
  - Research Site, Chula Vista, California
  - Research Site, Huntington Park, California
  - Research Site, Lincoln, California
  - Research Site, Los Angeles, California
  - Research Site, Panorama City, California
  - Research Site, San Diego, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Gainesville, Florida
  - Research Facility, Miami, Florida
  - Research Site, Orlando, Florida
  - Reseaarch Site, Pompano Beach, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Marrero, Louisiana
  - Research Site, Oxon Hill, Maryland
  - Research Site, Wyoming, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Berlin, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Great Neck, New York
  - Research Site, Hartsdale, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lampasas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waxahachie, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No